CLINICAL TRIAL: NCT07264985
Title: Gut Microbiota Changes in Breast Cancer Patients Treated With Pyrotinib and Correlation With Drug-Induced Diarrhea: An Observational Cohort Study
Brief Title: Gut Microbiota and Diarrhea in Breast Cancer Patients Receiving Pyrotinib
Status: Not yet recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Other Study IDs: LLHBCH2025YN-087
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Drug-Related Side Effects; Diarrhea
Keywords: Pyrotinib; Diarrhea; Gut Microbiota; HER2-Positive Breast Cancer; Microbiome; Drug Side Effect; Metagenomics; Observational Study
MeSH Terms: conditions — Breast Neoplasms; Diarrhea; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces: Fresh stool samples (approximately 5g per collection) will be collected from participants at specified time points during pyrotinib treatment (e.g., at 2 weeks and 4 weeks). These samples will be immediately stored at -80°C. Genomic DNA will be extracted from these samples for metagenomic sequencing to analyze the composition and function of the gut microbiota.
  Blood: Peripheral blood samples (5mL in EDTA tubes for plasma and 5mL in serum separator tubes) will be collected during patient follow-up visits. After processing (centrifugation and aliquoting), the resulting plasma and serum samples will be stored at -80°C. These samples are intended for subsequent analyses, such as measuring systemic inflammatory cytokine levels (e.g., by ELISA) and potentially for metabolomic profiling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diarrhea Group: This cohort consists of HER2-positive breast cancer patients receiving pyrotinib treatment who develop diarrhea (graded as ≥ Grade 1 according to CTCAE v5.0) during the observation period. Participants in this group will provide stool samples and clinical data for comparison with the non-diarrhea group. No study intervention is administered; all patients receive standard medical care.
- Non-Diarrhea Group: This cohort consists of HER2-positive breast cancer patients receiving pyrotinib treatment who do not develop diarrhea (Grade 0 according to CTCAE v5.0) during the observation period. Participants in this group will provide stool samples and clinical data, serving as a control for comparison with the diarrhea group. No study intervention is administered; all patients receive standard medical care.

SUMMARY:
Background:

Pyrotinib is an effective targeted drug for HER2-positive breast cancer, but it very frequently causes diarrhea, which can be severe enough to disrupt treatment and reduce patients' quality of life. The reason why some patients develop diarrhea while others do not is not well understood. Recent research suggests that the community of bacteria in the gut (gut microbiota) may play a key role in this side effect.

What is the purpose of this study? This is an observational study (Phase 1) that aims to understand the relationship between pyrotinib treatment, changes in gut bacteria, and the occurrence of diarrhea. The main goal is to compare the gut bacteria of patients who develop diarrhea while taking pyrotinib with those who do not. Researchers hope to identify specific bacteria that might protect against diarrhea, which could lead to new ways to prevent or treat this side effect in the future.

What will happen in the study? Patients with HER2-positive breast cancer who are being treated with pyrotinib will be invited to participate. They will be divided into two groups: those who experience diarrhea and those who do not. Participants will provide stool samples at specific time points (e.g., 2 and 4 weeks after starting pyrotinib). They will also allow researchers to collect information from their medical records about their clinical condition and diarrhea symptoms. No experimental intervention will be administered in this phase of the study; all patients will receive standard medical care.

Potential Benefits:

Participants will not receive any direct benefit from this observational phase of the study. However, the information gathered may help scientists better understand pyrotinib-induced diarrhea and develop future strategies to help other breast cancer patients manage this side effect more effectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years, regardless of gender.
2. Diagnosed with HER2-positive breast cancer and currently receiving pyrotinib treatment (either as monotherapy or in combination with endocrine therapy), with a treatment duration of ≥ 2 weeks.
3. Voluntarily agree to participate in this study and provide written informed consent.

Exclusion Criteria:

1. History of significant gastrointestinal diseases (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis, intestinal obstruction) or previous major gastrointestinal surgery.
2. Recent use (within 1 month) of antibiotics, probiotics, or traditional Chinese medicine intended to alter intestinal function.
3. Pregnant or lactating women.
4. Patients who refuse to provide informed consent or explicitly express unwillingness to participate. Patients found not meeting the inclusion criteria after enrollment will be discontinued from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18-75) diagnosed with HER2-positive breast cancer who are currently undergoing treatment with pyrotinib (either as monotherapy or in combination). This is a prospective observational cohort study where participants are not assigned to an intervention but are instead grouped based on the natural outcome of whether they develop drug-induced diarrhea during the observation period. This creates two primary cohorts for comparison: the 'Diarrhea Group' and the 'Non-Diarrhea Group'. All participants will continue their standard pyrotinib treatment and clinical care throughout the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in gut microbiota β-diversity between the Diarrhea group and the Non-diarrhea group. | Through study completion, an average of 6 months.
  Beta diversity (e.g., using UniFrac distance) of the gut microbiota will be compared between the two groups based on metagenomic sequencing data. A statistically significant difference (P < 0.05) is expected.
Identification of specific bacterial species enriched in the Non-diarrhea group. | Through study completion, an average of 6 months.
  Metagenomic sequencing data will be analyzed to identify bacterial species that are significantly more abundant in the Non-diarrhea group compared to the Diarrhea group, using statistical methods such as LEfSe (Linear Discriminant Analysis Effect Size) with a threshold of LDA Score > 2 and P < 0.05.

SECONDARY OUTCOMES:
Difference in gut microbiota α-diversity between groups. | Through study completion, an average of 6 months.
  Alpha diversity indices (e.g., Shannon index, Chao1 index) of the gut microbiota will be compared between the Diarrhea and Non-diarrhea groups.
Differences in metagenomic functional pathways between groups. | Through study completion, an average of 6 months.
  Metagenomic sequencing data will be annotated using databases like KEGG. The abundance of functional pathways (e.g., KEGG Level 2 or 3) will be compared between the two groups to identify differentially abundant metabolic or functional modules.
Differences in serum inflammatory cytokine levels between groups. | Through study completion, an average of 6 months.
  Levels of systemic inflammatory cytokines (e.g., IL-6, TNF-α, CRP) measured in serum samples by ELISA or other assays will be compared between the Diarrhea and Non-diarrhea groups.
Differences in serum metabolomic profiles between groups. | Through study completion, an average of 6 months.
  Metabolomic profiling of serum samples will be performed (e.g., by mass spectrometry). The metabolic profiles will be compared between the two groups to identify differentially abundant metabolites.

OTHER OUTCOMES:
Predictive potential of baseline gut microbiota for pyrotinib-induced diarrhea risk. | Through study completion, an average of 6 months.
  An exploratory analysis to assess whether the composition and features of the gut microbiota before starting pyrotinib treatment (baseline) can predict the subsequent risk of developing diarrhea during treatment. Metagenomic sequencing data from baseline stool samples will be used to build predictive models.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) collected in this study will not be made publicly available. The primary reasons are to protect patient privacy and confidentiality, as the dataset contains detailed genetic (metagenomic) and clinical information that could potentially be used to identify individuals. Furthermore, the data is integral to ongoing and future research by the investigative team, including the development of synthetic probiotics, which may involve intellectual property considerations.